CLINICAL TRIAL: NCT00960856
Title: A Four Arm, Single-Dose, Food Effect Evaluation With 105 mg Fenofibric Acid Tablets Administered in a Fasted State and Three Different Fed Conditions, Low-Fat/Low Calorie Meal, Standard Meal, and High-Fat/High Calorie Meal
Brief Title: Four Arm Food Effect Study of Fenofibric Acid Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Vice President, Branded Products and Medical Affairs, Mutual Pharmaceutical Company, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-028-07-1009
Record Dates: First submitted 2009-08-14; First posted 2009-08-18 (Estimated); Results first posted 2009-10-14 (Estimated); Last update posted 2009-10-20 (Estimated); Status verified 2009-10

CONDITIONS: Healthy
Keywords: pharmacokinetics
MeSH Terms: interventions — fenofibric acid; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fenofibric Acid 105 mg - Low-Fat Meal (Experimental): Fenofibric Acid 105 mg tablet administered 30 minutes after the initiation of a low-fat breakfast.
  Interventions: Drug: Fenofibric Acid 105 mg Tablet
- Fenofibric Acid 105 mg - Standard Meal (Experimental): Fenofibric Acid 105 mg tablet administered 30 minutes after the initiation of a standard breakfast.
  Interventions: Drug: Fenofibric Acid 105 mg Tablet
- Fenofibric Acid 105 mg - High-Fat/High-Calorie Meal (Experimental): Fenofibric Acid 105 mg tablet administered 30 minutes after the initiation of a high-fat/high-calorie breakfast.
  Interventions: Drug: Fenofibric Acid 105 mg Tablet
- Fenofibric Acid 105 mg - Fasted State (Experimental): Fenofibric Acid 105 mg tablet administered after an overnight fast of at least 10 hours
  Interventions: Drug: Fenofibric Acid 105 mg Tablet

INTERVENTIONS:
Drug: Fenofibric Acid 105 mg Tablet — One 105 mg tablet administered 30 minutes after the initiation of a low-fat breakfast.
  Arms: Fenofibric Acid 105 mg - Low-Fat Meal
Drug: Fenofibric Acid 105 mg Tablet — One 105 mg tablet administered 30 minutes after the initiation of a standard breakfast
  Arms: Fenofibric Acid 105 mg - Standard Meal
Drug: Fenofibric Acid 105 mg Tablet — One 105 mg tablet administered 30 minutes after the initiation of a high-fat/high-calorie breakfast.
  Arms: Fenofibric Acid 105 mg - High-Fat/High-Calorie Meal
Drug: Fenofibric Acid 105 mg Tablet — One 105 mg tablet administered after an overnight fast of at least 10 hours.
  Arms: Fenofibric Acid 105 mg - Fasted State

SUMMARY:
The primary objective of this study is to characterize the single-dose pharmacokinetic profile of fenofibric acid (105 mg tablets) and the effect of food of various calorie/fat compositions on the rate and extent of absorption. Additionally, the safety and tolerability of this dose and regimen of fenofibric acid will be evaluated.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the single-dose pharmacokinetic profile of fenofibric acid (105 mg tablets) and the effect of food of various calorie/fat compositions on the rate and extent of absorption. Forty healthy, non-smoking, non-obese, non-pregnant adult volunteers between the ages of 18 and 45 years old will receive a single oral dose of fenofibric acid in one of four randomly assigned sequences of meal conditions each separated by a 7 day washout period. On study Days 1, 8, 15 and 22 each subject will receive a single oral dose (1 x 105 mg tablet) of fenofibric acid following an overnight fast of at least 10 hours or with a low-fat meal, standard meal, or high-fat/high-calorie meal according to their randomization sequence. Subjects will fast for at least 4.25 hours after dosing in each of the four dosing conditions. Blood samples will be drawn from all participants before dosing and for 72 hours post-dose at times sufficient to adequately define the pharmacokinetics of fenofibric acid. A further goal of this study is to evaluate the safety and tolerability of this regimen in healthy volunteers. Seated blood pressure and heart rate will be measured prior to dosing and at 2 hours post-dose. Subjects will be monitored throughout the confinement portion of the study for adverse reactions to the study drug and/or procedures. All adverse events whether elicited by query, spontaneously reported, or observed by clinic staff will be evaluated by the Investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between the ages of 18 and 45
* Non-smoking
* Non-pregnant (post-menopausal, surgically sterile, or using effective contraceptive measures)
* Body mass index (BMI) less than 30
* Medically healthy on the basis of medical history and physical examination
* Hemoglobin > or = to 12g/dL
* Completion of the screening process within 28 days prior to dosing
* Provision of voluntary written informed consent

Exclusion Criteria:

* Recent participation (within 28 days) in other research studies
* Recent significant blood donation or plasma donation
* Pregnant or lactating
* Test positive at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV)
* Recent (2-year) history or evidence of alcoholism or drug abuse
* History or presence of significant cardiovascular, pulmonary, hepatic, gallbladder or biliary tract, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
* Subjects who have used any drugs or substances known to inhibit or induce cytochrome (CYP) P450 enzymes and/or P-glycoprotein (P-gp) within 28 days prior to the first dose and throughout the study
* Drug allergies to fenofibric acid

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2007-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PRACS Institute, Ltd. - Cetero Research, Fargo, North Dakota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Non-obese, non-smoking, healthy adult volunteers consisting of members of the community-at-large were enrolled.
Pre-assignment Details: 88 subjects were screened and 51 were screen failures. Enrollment of 40 subjects was planned, however, the enrollment of 37 subjects was judged to be sufficient to meet the criterion of 36 necessary to complete the study.
Groups:
- Sequence ABCD; Sequence BCDA; Sequence CDAB; Sequence DABC: Participants received one 105 mg fenofibric acid tablet following each of the following four meal conditions, in this order: A= Low-fat meal, B= standard meal, C= high-fat/high-calorie meal, D= fasted state.
Period: Period I
Arm/Group | Sequence ABCD | Sequence BCDA | Sequence CDAB | Sequence DABC
Started | 10 | 9 | 9 | 9
Completed | 10 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period of 7 Days
Arm/Group | Sequence ABCD | Sequence BCDA | Sequence CDAB | Sequence DABC
Started | 10 | 9 | 9 | 9
Completed | 10 | 7 (personal reasons) | 9 | 9
Not Completed | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0
Period: Period II
Arm/Group | Sequence ABCD | Sequence BCDA | Sequence CDAB | Sequence DABC
Started | 10 | 7 | 9 | 9
Completed | 10 | 7 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period of 7 Days
Arm/Group | Sequence ABCD | Sequence BCDA | Sequence CDAB | Sequence DABC
Started | 10 | 7 | 9 | 9
Completed | 10 | 7 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Period III
Arm/Group | Sequence ABCD | Sequence BCDA | Sequence CDAB | Sequence DABC
Started | 10 | 7 | 9 | 9
Completed | 10 | 7 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period of 7 Days
Arm/Group | Sequence ABCD | Sequence BCDA | Sequence CDAB | Sequence DABC
Started | 10 | 7 | 9 | 9
Completed | 10 | 7 | 8 | 9
Not Completed | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Period: Period IV
Arm/Group | Sequence ABCD | Sequence BCDA | Sequence CDAB | Sequence DABC
Started | 10 | 7 | 8 | 9
Completed | 10 | 7 | 8 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Low-Fat Meal, Standard Meal, High Fat/High Calorie Meal,Fasted: All subjects received each of the four study regimens in a randomly assigned sequence of dosing periods. On the mornings of Days 1, 8, 15 and 22 each subject received one tablet of fenofibric acid 105 mg administered after one of the following meal conditions: 1) low-fat meal, 2) standard meal, 3) high-fat/high-calorie meal 4) overnight fast of at least 10 hours.
Arm/Group | Low-Fat Meal, Standard Meal, High Fat/High Calorie Meal,Fasted
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 23.89 (6.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum or peak concentration that the drug reaches in the plasma.
Time Frame: serial pharmacokinetic blood samples drawn immediately prior to dosing and then 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours after dose administration
Population: Pharmacokinetic analyses of fenofibric acid are based on 34 subjects who completed the study. One subject discontinued due to an adverse event and two subjects discontinued for personal reasons.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Low-fat Meal - Treatment A: Each subject received one tablet of 105 mg fenofibric acid 30 minutes after the initiation of a low-fat breakfast.
- Standard Meal - Treatment B: Each subject received one tablet of 105 mg fenofibric acid 30 minutes after the initiation of a standard breakfast.
- High-Fat, High-Calorie Meal - Treatment C: Each subject received one tablet of 105 mg fenofibric acid 30 minutes after the initiation of a high-fat, high-calorie breakfast.
- Fasted - Treatment D: Each subject received one tablet of 105 mg fenofibric acid after an overnight fast of at least 10 hours.
Arm/Group | Low-fat Meal - Treatment A | Standard Meal - Treatment B | High-Fat, High-Calorie Meal - Treatment C | Fasted - Treatment D
Number analyzed (Participants) | 34 | 34 | 34 | 34
ng/mL | 9,806.74 (2,120.78) | 9,854.39 (1,980.77) | 7,950.75 (1,920.85) | 12,061.67 (2,241.31)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the plasma concentration versus time curve, from time 0 to the time of the last measurable concentration (t), as calculated by the linear trapezoidal rule.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Low-fat Meal - Treatment A | Standard Meal - Treatment B | High-Fat, High-Calorie Meal - Treatment C | Fasted - Treatment D
Number analyzed (Participants) | 34 | 34 | 34 | 34
ng-hr/mL | 132,636.84 (47,627.60) | 134,928.11 (50,262.64) | 134,814.42 (47,130.53) | 139,975.28 (48,821.99)

3. Primary Outcome: The Area Under the Plasma Concentration Versus Time Curve From Time 0 to Infinity AUC(0-∞)
Description: The area under the plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable plasma concentration to the elimination rate constant.
Time Frame: serial pharmacokinetic plasma concentrations were drawn prior to dose administration (0 hour) and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours after drug administration.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Low-fat Meal - Treatment A | Standard Meal - Treatment B | High-Fat, High-Calorie Meal - Treatment C | Fasted - Treatment D
Number analyzed (Participants) | 34 | 34 | 34 | 34
ng-hr/mL | 145,827.10 (56,137.08) | 148,367.21 (58,828.43) | 148,488.53 (55,949.04) | 152,571.61 (55,060.83)

ADVERSE EVENTS:
Description: 37 subjects were enrolled in this study. Several subjects dropped out of the study prior to receiving all interventions. 35 subjects were administered Fenofibric Acid 105 mg tablets with a low fat meal, high fat meal and in a fasted state. 36 subjects were administered Fenofibric Acid 105 mg tablets with a standard meal.
Groups:
- Fasted - Treatment D: Each subject received one tablet of 105 mg fenofibric acid following an overnight fast of at least 10 hours.
Arm/Group | Low-Fat Meal - Treatment A | Standard Meal - Treatment B | High-fat, High-calorie Meal - Treatment C | Fasted - Treatment D
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36 | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 9/35 | 2/36 | 4/35 | 4/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-Fat Meal - Treatment A (N=35) | Standard Meal - Treatment B (N=36) | High-fat, High-calorie Meal - Treatment C (N=35) | Fasted - Treatment D (N=35)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site hematoma (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Vessel puncture site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine kinase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days